CLINICAL TRIAL: NCT00827684
Title: Phase II Study of Temsirolimus and Irinotecan in Chemotherapy Refractory Patients With KRAS Mutated Metastatic Colorectal Cancer
Brief Title: Temsirolimus and Irinotecan for Treatment Resistant Patients With Metastatic Colorectal Cancer and KRAS Mutations
Acronym: TIRASMUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Professor, MD, DMSc Andes Jakobsen, Dept. of Oncology, Vejle Hospital
Purpose: Treatment
Other Study IDs: 2008-007665-22
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: KRAS mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Response or stable disease (Active Comparator): will receive Temsirolimus
  Interventions: Drug: Temsirolimus
- Progression (Experimental): Will receive a combination of Temsirolimus and Irinotecan
  Interventions: Drug: Irinotecan; Drug: Temsirolimus

INTERVENTIONS:
Drug: Irinotecan
  Arms: Progression
Drug: Temsirolimus

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of temsirolimus as a single drug, and of temsirolimus in combination with irinotecan in chemotherapy resistant patients with KRAS mutated colorectal cancer.

DETAILED DESCRIPTION:
Chemotherapy resistance is a major challenge in metastatic colorectal cancer (mCRC), and EGFR inhibitors have been introduced as 3rd line treatment to chemotherapy refractory patients. However, it has recently been established that response to treatment with irinotecan and cetuximab is confined to patients with wtKRAS tumors. Therefore, downstream targets are being proposed as potential inhibitors of the EGFR signalling in tumours with KRAS mutations. mTOR is a central intracellular signalling molecule and a rational approach for potential reversion of chemotherapy resistance in these patients.

Preclinical data suggest that different solid tumors could respond to mTOR inhibitors and report on enhanced antitumor activity in combination with different traditional cytostatic drugs. Furthermore recent preclinical data suggest that mTOR inhibition may induce tumor reduction in colon cancer xenographs. Temsirolimus (CCI-779) has been widely investigated in different clinical settings and is presently registered for treatment of renal cell carcinomas. Furthermore, is has recently shown response in metastatic breast cancer patients, but at present there are no clinical data on efficacy or safety in metastatic colorectal cancer patients.

The present study aims at investigating the safety and efficacy of monotherapy temsirolimus and a combination of temsirolimus and irinotecan in chemotherapy resistant, KRAS mutated colorectal adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified colorectal adenocarcinomas
* Age > 18 years and < 70
* Metastatic colorectal cancer refractory 5-FU, oxaliplatin and irinotecan containing treatment regimes
* KRAS mutation detected by DxS kit in primary tumor or metastatic lesion.
* Measurable disease according to RECIST
* ECOG performance status 0, 1 or 2
* Adequate renal, hepatic and haematological function
* Normal serum cholesterol and triglycerides
* Blood samples and available paraffin embedded tumor material for translational research studies
* Fertile males and females (< 2 years after last period for women) must use effective birth control
* Signed Informed consent

Exclusion Criteria:

* Clinically significant heart disease, active severe infections or other concurrent disease
* Other malignant diseases within 5 years of inclusion in the study, except basal cell squamous cell carcinoma of the skin and cervical carcinoma-in-situ
* Prior radiotherapy within 30 days of treatment start
* Other experimental therapy within 30 days of treatment initiation
* Patients who are breast feeding, childbearing or of childbearing potential without using dual effective contraception
* Clinical or radiological evidence of CNS metastasis
* Completed any major surgery, excision biopsy or significant traumatic lesion ≥ 4 weeks from start of treatment and completed any minor surgery ≥ 1 week prior to start of treatment

  * Insertion of a vascular access device is not considered major or minor surgery from the viewpoint of protocol eligibility
  * Patients must have fully recovered from the procedure and have a fully healed incision
* Planned radiation therapy against target-lesions
* Patients with significant non-healing wounds or ulcers
* History or evidence of thrombotic or hemorrhagic disorders

  * Significant haemorrhage (> 30 ml/bleeding episode in previous 3 months)
  * Haemoptysis (> 5 ml fresh blood in previous 4 weeks)
* Patients on full-dose anticoagulation (e.g., warfarin) are eligible provided that both of the following criteria are met:

  * The patient has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or is on a stable dose of low molecular weight heparin
  * The patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub-Arachnoid Hemorrhage (SAH) within 12 months prior to randomization
* No known or history of HIV seropositivity
* The use of ACE inhibitors is not permitted during the study
* Known allergy to temsirolimus, sirolimus, polysorbate 80 or included agents.
* Agents with strong CYP3A4-inhibitory potential

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Objective response rates

SECONDARY OUTCOMES:
Progression free survival
Overall survival
Translational Research

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, MD, DMSc, Study Chair — Vejle Hospital; Karen-Lise G Spindler, MD, PhD, Principal Investigator — Vejle Hospital
Locations (2):
- Denmark (2):
  - Rigshospitalet, Department of Oncology, Copenhagen
  - Vejle Hospital, Dept. of Oncology, Vejle